CLINICAL TRIAL: NCT05043220
Title: COVID-19-Prädiktoren: Klinische Studie Zur Sicherheit Von Gynäkologisch Onkologischen Patientinnen Unter Onkologischer Systemtherapie - CO-SI-ONKO-Studie
Brief Title: Covid-19 Predictors: Safety of Gynecological Oncology Patients Undergoing Systemic Cancer Therapy
Acronym: CO-SI-ONKO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Heike Jansen, Principal Investigator, Technical University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CO-SI-ONKO
Record Dates: First submitted 2021-09-13; First posted 2021-09-14 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Telemedicine (Experimental): Telemonitoring via PPG (photoplethysmography) and PROM (patient reported outcome monitoring) via app
  Interventions: Device: PPG and PROM

INTERVENTIONS:
Device: PPG and PROM — description will follow

SUMMARY:
We designed a monocenter prospective cohort study using PROM via app and remote monitoring via pho-toplethysmography (PPG). The application of these technologies enables an early detection of infections and therefore initiation of medical interventions. The study is conducted as feasibility analysis; primary endpoints are adherence (according to wearing time) and technical robustness.

ELIGIBILITY:
Inclusion Criteria:

* gynecological cancer
* indication for systemic cancer therapy
* patients who are legally competent and able to understand and follow instructions of the study staff
* present informed consent

Exclusion Criteria:

* no use if internet or applications
* persons who are in a dependency or employment relationship with the study center
* positive proof of COVID-19
* affection of the external auditory canal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Compliance | 3 months
  Compliance is defined as wearing time of the in-ear-sensor.
robustness of the ppg-signal | 3 months
  number and duration of the ppg-signal transmitted

SECONDARY OUTCOMES:
number of correct- and false-positive alerts | 3 months
  definition via comparison of alerts with clinical data
number of contacts and hospitalization rates | 3 months
  definition via comparison of alerts and resulting contacts and hospitalization rates with clinical data
infections | 3 months
  detection of infesctions via suspected ppg-signal transmitted or PRO-data. This results in blood test zu verify acute infections.
therapy modifications | 3 months
  dose-reductions (%), postponing of therapy cycles (time in days between actual and plannend date), therapy discontinuation
effect on quality of life | 3 months
  change in minimum 9 points in the EORTC QLQ-C30-questionnaire is evaluated as significant change. In questions 1-28: 28-112 points can be achieved: higher scores are associated with a worse outcome. In questions 29-30:2-14 points can be achieved: higher scores are associated with a better outcome.
OS; PFS | 3 months
  time between study inclusion and death; time between study inclusion and proven increasing tumor mass (number of days)
health-related costs | 3 months
  cost-effectiveness analysis

CONTACTS AND LOCATIONS:
Overall Officials: Heike Jansen, Dr. med, Principal Investigator — Technical University of Munich; Marion Kiechle, Prof. Dr. med., Study Director — Technical University of Munich
Locations (1):
- Klinikum rechts der Isar, Frauenklinik, Technische Universität München, Munich, Germany